CLINICAL TRIAL: NCT03467425
Title: The Clinical Effectiveness of Fluticasone Furoate/Umeclidinium Bromide/Vilanterol in a Single Inhaler (TRELEGY™ ELLIPTA™) When Compared With Non-ELLIPTA Multiple Inhaler Triple Therapies in COPD Patients Within a Usual Care Setting
Brief Title: INTREPID: Investigation of TRELEGY Effectiveness: Usual Practice Design
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 206854; 2017-004369-29 (EudraCT Number)
Record Dates: First submitted 2018-02-02; First posted 2018-03-16 (Actual); Results first posted 2020-09-07 (Actual); Last update posted 2020-09-07 (Actual); Status verified 2020-07

CONDITIONS: Pulmonary Disease, Chronic Obstructive
Keywords: FF/VI/UMEC; TRELEGY ELLIPTA; COPD; Effectiveness
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Intervention Model Description: Subjects will be randomized in a ratio of 1:1 to receive one of the following study treatment regimens: TRELEGY ELLIPTA once daily in the morning or Non-ELLIPTA MITT twice-daily treatment.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- TRELEGY ELLIPTA (FF/UMEC/VI: 100 mcg/62.5 mcg/25 mcg) (Experimental): Eligible subjects will receive a blended combination of FF in the first strip (100 mcg per blister) and UMEC/VI in second strip (62.5 mcg UMEC per blister and 25 mcg VI per blister), a single inhalation once daily in the morning in the same TRELEGY ELLIPTA Dry Powder Inhaler (DPI) via inhalation route for a period of 24 weeks. Study treatment may be augmented with other prescribed COPD medications such as including rescue medications, which will be prescribed and obtained according to usual practice.
  Interventions: Drug: FF/UMEC/VI; Drug: COPD rescue medications
- Non-ELLIPTA MITT (Active Comparator): Eligible subjects will receive the ICS/LAMA/LABA products twice daily and dosing regimens as prescribed by their physician for a period of 24 weeks. Study treatment may be augmented with other prescribed COPD medications such as including rescue medications, which will be prescribed and obtained according to usual practice.
  Interventions: Drug: Inhaled Corticosteroid; Drug: LAMA; Drug: LABA; Drug: COPD rescue medications

INTERVENTIONS:
Drug: FF/UMEC/VI — FF is a dry white powder containing 100 mcg GW685698 blended with lactose in one blister in the first strip of the DPI. UMEC/VI is a dry white powder containing 62.5 mcg of UMEC and 25 mcg of VI per blister, both blended together with lactose and magnesium stearate in the second strip of the DPI.
  Arms: TRELEGY ELLIPTA (FF/UMEC/VI: 100 mcg/62.5 mcg/25 mcg)
Drug: Inhaled Corticosteroid — Inhaled Corticosteroid (ICS) as prescribed by the physician.
  Arms: Non-ELLIPTA MITT
Drug: LAMA — LAMA as prescribed by the physician.
  Arms: Non-ELLIPTA MITT
Drug: LABA — LABA as prescribed by the physician.
  Arms: Non-ELLIPTA MITT
Drug: COPD rescue medications — Rescue medications for COPD will be prescribed and obtained according to usual practice.

SUMMARY:
The primary purpose of this study is to assess the effectiveness of TRELEGY ELLIPTA relative to non-ELLIPTA Multiple Inhaler Triple Therapies (MITT) for Chronic Obstructive Pulmonary Disease (COPD) control within the usual clinical practice setting. The study will be conducted once TRELEGY ELLIPTA has been approved in the countries in which the study will be conducted and is available commercially. This is a randomized, open-label, effectiveness, phase 4 study of 24 weeks' duration in COPD subjects to evaluate TRELEGY ELLIPTA (fluticasone furoate [FF]/vilanterol [VI]/umeclidinium bromide [UMEC]: 100 microgram [mcg]/62.5 mcg/25 mcg) inhalation powder taken once daily using a single ELLIPTA inhaler compared with any non-ELLIPTA MITT in the usual care setting. Effectiveness of TRELEGY ELLIPTA will be assessed by comparing proportion of COPD Assessment Test (CAT) responders at Week 24 between two treatment groups. TRELEGY and ELLIPTA are trademarks of GlaxoSmithKline (GSK) group of companies. The study will enroll approximately 3000 subjects.

ELIGIBILITY:
Inclusion Criteria:

* Capable of giving signed informed consent.
* Subjects with a documented physician diagnosis of COPD.
* A score of >=10 on the CAT at screening.
* Subjects who have a history of treatment with systemic/oral corticosteroids, antibiotics and/or hospitalization for at least one COPD exacerbation in the 3 years prior to randomization. This will be captured through subject recall and/or medical records and must be documented in subject's notes. Prior use of systemic/oral corticosteroids and/or antibiotics alone does not qualify as an exacerbation history unless the use was associated with treatment of worsening symptoms of COPD.
* Subjects currently receiving one of the non-ELLIPTA maintenance therapies listed below who have been prescribed it continually for at least 16 weeks prior to randomization. Continuous prescription is defined as a minimum of 60 days' prescription cover during the prior 16 weeks. The non-ELLIPTA maintenance therapy must be one of the following: Inhaled Corticosteroid (ICS) in combination with Long-acting Muscarinic Receptor Antagonist (LAMA) and Long Acting Beta-Agonist (LABA) (MITT) or LAMA and LABA used in combination as a dual therapy or LABA and ICS used in combination as a dual therapy. Subjects who are currently on a dual maintenance therapy for COPD must be considered by their physician to require a step-up to triple therapy. The reason for the physician decision to step- up must be documented. Subjects who are receiving only COPD medication on an 'as required' basis are not eligible.
* Subjects must be aged >=40 years of age at the time of signing the informed consent.

Exclusion Criteria:

* Women of child bearing potential: Women who are pregnant or lactating or are planning on becoming pregnant during the study.
* Subjects with any life-threatening condition i.e. low probability, in the opinion of the investigator, of 6-month survival due to severity of COPD or comorbid condition.
* Subjects with resolution of an exacerbation less than 2 weeks prior to visit 1, must not be randomized. Subjects may be rescreened 2 weeks after resolution of exacerbation (exacerbation is defined by treatment with systemic corticosteroids and/or antibiotic).
* Subjects with historical or current evidence of uncontrolled or clinically significant disease. Significant is defined as any disease that, in the opinion of the investigator, would put the safety of the subject at risk through participation, or which would affect the effectiveness or safety analysis if the disease/condition exacerbated during the study.
* A history of allergy or hypersensitivity to any corticosteroid, anticholinergic/muscarinic receptor antagonist, beta2-agonist, lactose/milk protein or magnesium stearate or a medical condition such as narrow-angle glaucoma, prostatic hypertrophy or bladder neck obstruction that, in the opinion of the investigator contraindicates study participation.
* Subjects who, in the opinion of the treating investigator, are chronic users of oral corticosteroids for respiratory or other indications (if unsure discuss with the medical monitor prior to screening). Chronic use is defined as more than 14 days continuous use during the 12 weeks prior to visit 1.
* Subjects taking any investigational drug treatment within 30 days prior to Visit 1 or within five half-lives (t½) of the prior investigational study (whichever is the longer of the two).

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3109 (Actual)
Dates: Start 2018-04-11 (Actual); Primary Completion 2019-10-10 (Actual); Study Completion 2019-10-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (116):
- Germany (36):
  - GSK Investigational Site, Aschaffenburg, Bavaria
  - GSK Investigational Site, Dachau, Bavaria
  - GSK Investigational Site, Garmisch-Partenirchen, Bavaria
  - GSK Investigational Site, Wallerfing, Bavaria
  - GSK Investigational Site, Cottbus, Brandenburg
  - GSK Investigational Site, Fürstenwalde, Brandenburg
  - GSK Investigational Site, Potsdam, Brandenburg
  - GSK Investigational Site, Rüdersdorf, Brandenburg
  - GSK Investigational Site, Darmstadt, Hesse
  - GSK Investigational Site, Frankfurt am Main, Hesse
  - GSK Investigational Site, Fulda, Hesse
  - GSK Investigational Site, Marburg, Hesse
  - GSK Investigational Site, Rodgau, Hesse
  - GSK Investigational Site, Rüsselsheim am Main, Hesse
  - GSK Investigational Site, Hanover, Lower Saxony
  - GSK Investigational Site, Peine, Lower Saxony
  - GSK Investigational Site, Wardenburg, Lower Saxony
  - GSK Investigational Site, Bergisch Gladbach, North Rhine-Westphalia
  - GSK Investigational Site, Bonn, North Rhine-Westphalia
  - GSK Investigational Site, Cologne, North Rhine-Westphalia
  - GSK Investigational Site, Essen, North Rhine-Westphalia
  - GSK Investigational Site, Gelsenkirchen, North Rhine-Westphalia
  - GSK Investigational Site, Rheine, North Rhine-Westphalia
  - GSK Investigational Site, Warendorf, North Rhine-Westphalia
  - GSK Investigational Site, Koblenz, Rhineland-Palatinate
  - GSK Investigational Site, Delitzsch, Saxony
  - GSK Investigational Site, Leipzig, Saxony
  - GSK Investigational Site, Halle, Saxony-Anhalt
  - GSK Investigational Site, Teuchern, Saxony-Anhalt
  - GSK Investigational Site, Geesthacht, Schleswig-Holstein
  - GSK Investigational Site, Lübeck, Schleswig-Holstein
  - GSK Investigational Site, Schleswig, Schleswig-Holstein
  - GSK Investigational Site, Schmölln, Thuringia
  - GSK Investigational Site, Berlin
  - GSK Investigational Site, Deggendorf
  - GSK Investigational Site, Hamburg
- Netherlands (13):
  - GSK Investigational Site, Alkmaar
  - GSK Investigational Site, Breda
  - GSK Investigational Site, Dordrecht
  - GSK Investigational Site, Groningen
  - GSK Investigational Site, Harderwijk
  - GSK Investigational Site, Heerlen
  - GSK Investigational Site, Hengelo
  - GSK Investigational Site, Hoorn
  - GSK Investigational Site, Kloosterhaar
  - GSK Investigational Site, Nijmegen
  - GSK Investigational Site, Rotterdam
  - GSK Investigational Site, Zeist
  - GSK Investigational Site, Zutphen
- Spain (22):
  - GSK Investigational Site, Marbella - Málaga, Andalusia
  - GSK Investigational Site, Laredo, Cantabria
  - GSK Investigational Site, Torrejón de Ardoz, Madrid
  - GSK Investigational Site, Alcorcón (Madrid)
  - GSK Investigational Site, Alzira/Valencia
  - GSK Investigational Site, Barcelona
  - GSK Investigational Site, Basurto/Bilbao
  - GSK Investigational Site, Benalmádena, Málaga
  - GSK Investigational Site, Cadiz
  - GSK Investigational Site, Cáceres
  - GSK Investigational Site, L'Hospitalet de Llobregat. Barcelona
  - GSK Investigational Site, La Roca Del Valles (Barcelona)
  - GSK Investigational Site, Logroño
  - GSK Investigational Site, Loja/ Granada
  - GSK Investigational Site, Madrid
  - GSK Investigational Site, Palma de Mallorca
  - GSK Investigational Site, Ponferrada (León)
  - GSK Investigational Site, Pozuelo de Alarcón/Madrid
  - GSK Investigational Site, Segovia
  - GSK Investigational Site, Seville
  - GSK Investigational Site, Vigo-Pontevedra
  - GSK Investigational Site, Zaragoza
- Sweden (15):
  - GSK Investigational Site, Angered
  - GSK Investigational Site, Flen
  - GSK Investigational Site, Gothenburg
  - GSK Investigational Site, Härnösand
  - GSK Investigational Site, Höllviken
  - GSK Investigational Site, Kristianstad
  - GSK Investigational Site, Kungsbacka
  - GSK Investigational Site, Luleå
  - GSK Investigational Site, Malmo
  - GSK Investigational Site, Motala
  - GSK Investigational Site, Örebro
  - GSK Investigational Site, Östersund
  - GSK Investigational Site, Södertälje
  - GSK Investigational Site, Stockholm
  - GSK Investigational Site, Trollhättan
- United Kingdom (30):
  - GSK Investigational Site, Soham, Cambridgeshire
  - GSK Investigational Site, Llanelli, Carmarthenshire
  - GSK Investigational Site, Bollington, Cheshire
  - GSK Investigational Site, Macclesfield, Cheshire
  - GSK Investigational Site, Sandbach, Cheshire
  - GSK Investigational Site, Rhyl, Denbighshire
  - GSK Investigational Site, Waterlooville, Hampshire
  - GSK Investigational Site, Wishaw, Lanarkshire
  - GSK Investigational Site, Corby, Northamptonshire
  - GSK Investigational Site, Wellingborough, Northamptonshire
  - GSK Investigational Site, Leiston, Suffolk
  - GSK Investigational Site, Bexhill-on-Sea, Sussex East
  - GSK Investigational Site, Gateshead, Tyne & Wear
  - GSK Investigational Site, Bebington
  - GSK Investigational Site, Buckley
  - GSK Investigational Site, Cardiff
  - GSK Investigational Site, Colchester
  - GSK Investigational Site, Corbridge
  - GSK Investigational Site, Cornwall
  - GSK Investigational Site, Edinburgh
  - GSK Investigational Site, Hull
  - GSK Investigational Site, Irlam, Manchester
  - GSK Investigational Site, Larbet
  - GSK Investigational Site, Manchester
  - GSK Investigational Site, Newport
  - GSK Investigational Site, Newport, Isle of Wight
  - GSK Investigational Site, Poole
  - GSK Investigational Site, Southampton
  - GSK Investigational Site, Swinton
  - GSK Investigational Site, Warrington

IPD SHARING:
Plan to Share IPD: Yes
IPD for this study will be made available via the Clinical Study Data Request site.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: IPD will be made available within 6 months of publishing the results of the primary endpoints of the study.
Access Criteria: Access is provided after a research proposal is submitted and has received approval from the Independent Review Panel and after a Data Sharing Agreement is in place. Access is provided for an initial period of 12 months but an extension can be granted, when justified, for up to another 12 months.
URL: http://clinicalstudydatarequest.com

REFERENCES:
- [Derived] Worsley S, Snowise N, Halpin DMG, Midwinter D, Ismaila AS, Irving E, Sansbury L, Tabberer M, Leather D, Compton C. Clinical effectiveness of once-daily fluticasone furoate/umeclidinium/vilanterol in usual practice: the COPD INTREPID study design. ERJ Open Res. 2019 Nov 4;5(4):00061-2019. doi: 10.1183/23120541.00061-2019. eCollection 2019 Oct. PMID 31720293

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This was a Phase IV, open-label, randomized study to evaluate the effectiveness of TRELEGY ELLIPTA relative to non-ELLIPTA multiple inhaler triple therapies (MITT) for chronic obstructive pulmonary disease (COPD) control within the usual clinical practice setting. TRELEGY and ELLIPTA are registered trademarks of GlaxoSmithKline group of companies.
Pre-assignment Details: A total of 3341 participants were screened and 3109 participants (Par.) were enrolled in this study. Of which, 3092 participants were randomized and received the study treatment. The remaining 17 participants were randomized in error (those who were recorded as screen failures and also randomized) and did not receive investigational product (IP).
Groups:
- FF /UMEC/VI: 100 mcg/62.5 mcg/25 mcg by ELLIPTA DPI: Eligible participants received a combination of fluticasone furoate (FF) blended with lactose in the first strip (100 microgram [mcg] per blister); and umeclidinium bromide (UMEC) and vilanterol (VI) blended with lactose and magnesium stearate in second strip (62.5 mcg UMEC per blister and 25 mcg VI per blister), a single inhalation once daily in the same TRELEGY ELLIPTA dry powder inhaler (DPI) via inhalation route for a period of 24 weeks. Participants were administered other prescribed COPD medications such as rescue medications according to usual practice, as suggested by physician.
- Non-ELLIPTA MITT: Eligible participants received the inhaled corticosteroid (ICS)/long-acting muscarinic receptor antagonist (LAMA)/long-acting beta agonist (LABA) products twice daily as prescribed by the physician for a period of 24 weeks. Participants were administered other prescribed COPD medications such as rescue medications according to usual practice, as suggested by physician.
Period: Overall Study
Arm/Group | FF /UMEC/VI: 100 mcg/62.5 mcg/25 mcg by ELLIPTA DPI | Non-ELLIPTA MITT
Started | 1545 | 1547
Randomized But Did Not Start IP | 1 | 0
Completed IP | 1256 | 1359
Not Completed IP | 288 | 188
Withdrew IP (WIP): Lost to Follow-up | 15 | 24
WIP: Protocol Deviation | 0 | 2
WIP: Adverse Event | 112 | 29
WIP: Lack of Efficacy | 56 | 28
WIP: Physician Decision | 14 | 27
WIP: Withdrawal by Participant | 91 | 78
Completed | 1498 | 1493
Not Completed | 47 | 54
Not completed — Adverse Event | 9 | 9
Not completed — Lack of Efficacy | 3 | 1
Not completed — Protocol Violation | 0 | 1
Not completed — Lost to Follow-up | 18 | 25
Not completed — Physician Decision | 2 | 1
Not completed — Withdrawal by Subject | 15 | 17

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | FF /UMEC/VI: 100 mcg/62.5 mcg/25 mcg by ELLIPTA DPI | Non-ELLIPTA MITT | Total
Number analyzed (Participants) | 1545 | 1547 | 3092
Age, Continuous [Mean (Standard Deviation); unit: Years] | 67.8 (8.78) | 67.8 (8.59) | 67.8 (8.68)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 708 | 729 | 1437
  Male | 837 | 818 | 1655
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Asian- Central/South Asian Heritage | 12 | 7 | 19
  Asian- East Asian Heritage | 0 | 1 | 1
  Asian- South East Asian Heritage | 1 | 6 | 7
  Black or African American | 3 | 4 | 7
  White- Arabic/North African Heritage | 6 | 7 | 13
  White- White/Caucasian/European Heritage | 1523 | 1521 | 3044
  White and Black or African American | 0 | 1 | 1

OUTCOME MEASURES:

1. Primary Outcome: Number of Responders and Non-responders Based on the Chronic Obstructive Pulmonary Disease Assessment Test (CAT) at Week 24 and Number of Participants With Imputed CAT Score at Week 24
Description: The CAT is a 8-item questionnaire, used to measure the health status of par. with COPD. Par. rated their experience on a 6-point scale: 0 (no impact) to 5 (maximum impact). CAT score was calculated by summing the non-missing scores of the 8 items with a range of 0-40. Higher scores indicate greater disease impact. Responders were par. who had a change from Baseline score >=2 at Week 24. Non-responders were the par. who had change from Baseline score <2 at Week 24. Change from Baseline was calculated as Week 24 value minus the Baseline value (Day 1). A composite strategy was applied when intercurrent events of randomized treatment modification, change in pulmonary rehabilitation or start of oxygen therapy occurred, otherwise a treatment policy strategy was applied. Missing Week 24 CAT data were imputed assuming missing at random and are presented in a separate category. Number of responders, non-responders based on CAT and par. with imputed CAT score at Week 24 are presented.
Time Frame: At Week 24
Population: Intent-to-Treat (ITT) Population comprised of all randomized participants (any participant who received a randomization number), excluding those who were randomized in error (a screen failure and also randomized). Only those participants with non-missing covariates were included in the analysis
Measure: Count of Participants; unit: Participants
Arm/Group | FF /UMEC/VI: 100 mcg/62.5 mcg/25 mcg by ELLIPTA DPI | Non-ELLIPTA MITT
Number analyzed (Participants) | 1539 | 1543
Participants
  Responders | 731 | 616
  Non-responders | 756 | 835
  Participants with imputed CAT score | 52 | 92
Statistical Analysis 1: Comparison: FF /UMEC/VI: 100 mcg/62.5 mcg/25 mcg by ELLIPTA DPI vs Non-ELLIPTA MITT; Test type: Superiority; p < 0.001, Regression, Logistic — Analysis was performed using logistic regression model with covariates of treatment group, Baseline CAT score, number of exacerbations in the prior year, actual prior medication use strata and country; Odds Ratio (OR) = 1.31, 95% CI 2-sided [1.13 to 1.51] — Statistical comparison is presented for combined data of responders, non-responders and those with imputed CAT score at Week 24

2. Secondary Outcome: Change From Baseline in Forced Expiratory Volume in 1 Second (FEV1) at Week 24
Description: FEV1 is a measure of lung function and is defined as the maximal amount of air that can be forcefully exhaled in one second. FEV1 measurements were collected using a spirometer. Baseline was defined as the value recorded at Day 1. Change from Baseline was calculated as FEV1 value at Week 24 minus the Baseline value. A treatment policy strategy was used for the intercurrent events of randomized treatment discontinuation, randomized treatment modification, change of pulmonary rehabilitation status and start of oxygen therapy. Only those participants with non-missing covariates were included in the analysis.
Time Frame: Baseline (Day 1) and at Week 24
Population: FEV1 Population comprised of all participants of the ITT population for whom a spirometry assessment was performed at any of Visit 1 (Day 1) or Visit 2 (Week 24). Only those participants with data available at the specified data points were analyzed.
Measure: Least Squares Mean (Standard Error); unit: Liters
Arm/Group | FF /UMEC/VI: 100 mcg/62.5 mcg/25 mcg by ELLIPTA DPI | Non-ELLIPTA MITT
Number analyzed (Participants) | 691 | 675
Liters | 1.446 (0.0105) | 1.396 (0.0108)
Statistical Analysis 1: Comparison: FF /UMEC/VI: 100 mcg/62.5 mcg/25 mcg by ELLIPTA DPI vs Non-ELLIPTA MITT; Test type: Superiority; p < 0.001, ANCOVA; Mean Difference (Net) = 0.050, 95% CI 2-sided [0.026 to 0.073], Standard Error of Mean 0.0121 — Analysis was performed using an ANCOVA with covariates of treatment group, Baseline FEV1, actual prior medication use strata, country and timing of spirometry

3. Secondary Outcome: Percentage of Participants Making at Least 1 Critical Error in Inhalation Technique at Week 24
Description: Participants were trained on the correct use of their inhaler devices. All participants who had spirometry measured were to have an assessment of inhaler errors. During the assessment, participants were asked to demonstrate inhaler use when taking their regular dose of medication. A critical error is defined as an error that is most likely to result in no or significantly reduced medication being inhaled. These errors were recorded in an error checklist, during the assessment. A hypothetical strategy was used for the intercurrent event of randomized treatment modification. Percentage of participants making at least 1 critical error in inhalation technique at the Week 24 is presented.
Time Frame: At Week 24
Population: Critical error Population comprised of all participants of the ITT population for whom a critical error assessment was performed at Visit 2 (Week 24). Only those participants with data available at the specified data points were analyzed.
Measure: Number; unit: Percentage of Participants
Arm/Group | FF /UMEC/VI: 100 mcg/62.5 mcg/25 mcg by ELLIPTA DPI | Non-ELLIPTA MITT
Number analyzed (Participants) | 653 | 230
Percentage of Participants | 6 | 3
Statistical Analysis 1: Comparison: FF /UMEC/VI: 100 mcg/62.5 mcg/25 mcg by ELLIPTA DPI vs Non-ELLIPTA MITT; Test type: Superiority; p = 0.103, Regression, Logistic; Odds Ratio (OR) = 1.99, 95% CI 2-sided [0.87 to 4.53] — Analysis was performed using logistic regression model with covariates of treatment group, actual prior medication use strata and country

ADVERSE EVENTS:
Time Frame: Serious adverse events (SAEs) and non-serious AEs (non-SAEs) were collected from the start of study treatment up to Week 24
Description: Data is reported for the ITT Population which comprised of all randomized participants (who received a randomization number), excluding those who were randomized in error. All SAEs were collected. Non-SAEs which were only drug-related or that lead to withdrawal from study/study treatment were collected.
Arm/Group | FF /UMEC/VI: 100 mcg/62.5 mcg/25 mcg by ELLIPTA DPI | Non-Ellipta MITT
All-Cause Mortality (participants affected / at risk) | 8/1545 | 8/1547
Serious Adverse Events (participants affected / at risk) | 114/1545 | 114/1547
Other Adverse Events (participants affected / at risk) | 32/1545 | 3/1547
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | FF /UMEC/VI: 100 mcg/62.5 mcg/25 mcg by ELLIPTA DPI (N=1545) | Non-Ellipta MITT (N=1547)
Pneumonia (Infections and infestations) | 26 (27) | 30 (30)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 26 (28) | 28 (29)
Infective exacerbation of chronic obstructive airways disease (Infections and infestations) | 6 (6) | 9 (9)
Acute myocardial infarction (Cardiac disorders) | 5 (5) | 5 (5)
Cardiac failure (Cardiac disorders) | 3 (3) | 7 (7)
Atrial fibrillation (Cardiac disorders) | 4 (4) | 5 (5)
Myocardial infarction (Cardiac disorders) | 5 (5) | 2 (2)
Fall (Injury, poisoning and procedural complications) | 2 (2) | 3 (3)
Sepsis (Infections and infestations) | 3 (3) | 2 (2)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 4 (4)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 3 (4) | 1 (1)
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 2 (2)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (2)
Humerus fracture (Injury, poisoning and procedural complications) | 2 (2) | 1 (1)
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 2 (2)
Peripheral arterial occlusive disease (Vascular disorders) | 2 (2) | 1 (1)
Peripheral ischaemia (Vascular disorders) | 1 (1) | 2 (2)
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 2 (2)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 0 (0)
Acute coronary syndrome (Cardiac disorders) | 1 (1) | 1 (1)
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2)
Angina pectoris (Cardiac disorders) | 2 (2) | 0 (0)
Ankle fracture (Injury, poisoning and procedural complications) | 2 (2) | 0 (0)
Cellulitis (Infections and infestations) | 2 (2) | 0 (0)
Cerebrovascular accident (Nervous system disorders) | 1 (1) | 1 (1)
Chest pain (General disorders) | 0 (0) | 2 (2)
Coronary artery disease (Cardiac disorders) | 1 (1) | 1 (1)
Diverticulum intestinal (Gastrointestinal disorders) | 1 (1) | 1 (1)
Femoral neck fracture (Injury, poisoning and procedural complications) | 0 (0) | 2 (2)
Femur fracture (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Hypertensive crisis (Vascular disorders) | 2 (2) | 0 (0)
Non-cardiac chest pain (General disorders) | 0 (0) | 2 (2)
Oesophageal carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1)
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Renal failure (Renal and urinary disorders) | 0 (0) | 2 (2)
Small cell lung cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1)
Syncope (Nervous system disorders) | 1 (1) | 1 (1)
Urosepsis (Infections and infestations) | 1 (1) | 1 (1)
Alcohol poisoning (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Anaemia (Blood and lymphatic system disorders) | 0 (0) | 1 (2)
Aortic valve stenosis (Cardiac disorders) | 1 (1) | 0 (0)
Atrial flutter (Cardiac disorders) | 0 (0) | 1 (1)
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Bladder perforation (Renal and urinary disorders) | 0 (0) | 1 (1)
Blood glucose increased (Investigations) | 0 (0) | 1 (1)
Brain stem infarction (Nervous system disorders) | 1 (1) | 0 (0)
Breast cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Cardiac arrest (Cardiac disorders) | 0 (0) | 1 (1)
Cardiac asthma (Cardiac disorders) | 1 (1) | 0 (0)
Cardiac failure chronic (Cardiac disorders) | 0 (0) | 1 (1)
Cardiogenic shock (Cardiac disorders) | 1 (1) | 0 (0)
Cerebral venous thrombosis (Nervous system disorders) | 1 (1) | 0 (0)
Cholecystitis (Hepatobiliary disorders) | 1 (1) | 0 (0)
Colitis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Constipation (Gastrointestinal disorders) | 0 (0) | 1 (1)
Cor pulmonale (Cardiac disorders) | 1 (1) | 0 (0)
Corynebacterium infection (Infections and infestations) | 0 (0) | 1 (1)
Death (General disorders) | 1 (1) | 0 (0)
Deep vein thrombosis (Vascular disorders) | 0 (0) | 1 (1)
Diplopia (Eye disorders) | 0 (0) | 1 (1)
Dizziness (Nervous system disorders) | 0 (0) | 1 (1)
Duodenal ulcer (Gastrointestinal disorders) | 1 (1) | 0 (0)
Dysuria (Renal and urinary disorders) | 1 (1) | 0 (0)
Enterocolitis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Erysipelas (Infections and infestations) | 1 (1) | 0 (0)
Fluid retention (Metabolism and nutrition disorders) | 0 (0) | 1 (2)
Gastrointestinal polyp haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1)
Gastrointestinal viral infection (Infections and infestations) | 1 (1) | 0 (0)
General physical health deterioration (General disorders) | 1 (1) | 0 (0)
Haemophilus infection (Infections and infestations) | 0 (0) | 1 (1)
Hodgkin's disease (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Hypersensitivity (Immune system disorders) | 1 (1) | 0 (0)
Hypokalaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hypomagnesaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hyponatraemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Iliac artery occlusion (Vascular disorders) | 1 (1) | 0 (0)
Incarcerated umbilical hernia (Gastrointestinal disorders) | 1 (1) | 0 (0)
Influenza (Infections and infestations) | 1 (1) | 0 (0)
Injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Large intestine perforation (Gastrointestinal disorders) | 1 (1) | 0 (0)
Large intestine polyp (Gastrointestinal disorders) | 0 (0) | 1 (1)
Left ventricular failure (Cardiac disorders) | 1 (1) | 0 (0)
Lower respiratory tract infection (Infections and infestations) | 0 (0) | 1 (1)
Lung squamous cell carcinoma stage II (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Mesothelioma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Multiple organ dysfunction syndrome (General disorders) | 1 (1) | 0 (0)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Necrotising fasciitis (Infections and infestations) | 0 (0) | 1 (1)
Nephrolithiasis (Renal and urinary disorders) | 0 (0) | 1 (1)
Non-small cell lung cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Osteolysis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Overdose (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Pancreatic carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Pancreatitis acute (Gastrointestinal disorders) | 1 (1) | 0 (0)
Peripheral artery occlusion (Vascular disorders) | 1 (1) | 0 (0)
Peroneal nerve palsy (Nervous system disorders) | 0 (0) | 1 (1)
Pituitary tumour benign (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Pleural mesothelioma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pneumonia haemophilus (Infections and infestations) | 1 (1) | 0 (0)
Pneumonia pneumococcal (Infections and infestations) | 0 (0) | 1 (1)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Presyncope (Nervous system disorders) | 1 (1) | 0 (0)
Pyelonephritis (Infections and infestations) | 0 (0) | 1 (1)
Rectal haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (2)
Respiratory syncytial virus bronchiolitis (Infections and infestations) | 1 (1) | 0 (0)
Respiratory tract infection (Infections and infestations) | 0 (0) | 1 (1)
Reversible ischaemic neurological deficit (Nervous system disorders) | 1 (1) | 0 (0)
Rhabdomyolysis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Rib fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Sensory loss (Nervous system disorders) | 0 (0) | 1 (1)
Shock haemorrhagic (Vascular disorders) | 1 (1) | 0 (0)
Shock hypoglycaemic (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Skin laceration (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Small cell lung cancer limited stage (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Small intestinal haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0)
Spinal fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Sudden death (General disorders) | 1 (1) | 0 (0)
T-cell lymphoma stage IV (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Toxicity to various agents (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Urinary bladder abscess (Infections and infestations) | 1 (1) | 0 (0)
Urinary tract infection (Infections and infestations) | 0 (0) | 1 (1)
Varicose vein (Vascular disorders) | 0 (0) | 1 (1)
Ventricular hypokinesia (Cardiac disorders) | 0 (0) | 1 (1)
Ventricular tachycardia (Cardiac disorders) | 1 (1) | 0 (0)
Vestibular disorder (Ear and labyrinth disorders) | 1 (1) | 0 (0)
Wound (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | FF /UMEC/VI: 100 mcg/62.5 mcg/25 mcg by ELLIPTA DPI (N=1545) | Non-Ellipta MITT (N=1547)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 32 (32) | 3 (3)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.

DOCUMENTS (2):
  • Study Protocol (2018-09-28): https://cdn.clinicaltrials.gov/large-docs/25/NCT03467425/Prot_000.pdf
  • Statistical Analysis Plan (2019-10-30): https://cdn.clinicaltrials.gov/large-docs/25/NCT03467425/SAP_001.pdf